CLINICAL TRIAL: NCT00646282
Title: Mineral Metabolism and Vascular Effects of Vitamin D Therapy in Kidney
Brief Title: Mineral Metabolism and Vascular Effects of Vitamin D Therapy in Kidney Transplant Patients
Acronym: PAD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment and discontinued once original principal investigator left Emory
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Antonio Guasch, M.D., Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006614
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Hyperparathyroidism, Secondary
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — 1 alpha-hydroxyergocalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doxercalciferol (Experimental): Stable kidney transplant recipients will receive Doxercalciferol
  Interventions: Drug: doxercalciferol
- Control (No Intervention): Stable kidney transplant recipients will not receive any drug

INTERVENTIONS:
Drug: doxercalciferol — The study drug dosage will be initiated according to baseline iPTH levels. For patients with iPTH>300 pg/ml, oral Doxercalciferol will be given at 1 mcg/day; for patients with iPTH <300 pg/ml, oral Doxercalciferol will be initiated at 0.5 mcg/day.
  Other Names: Hectorol
  Arms: Doxercalciferol

SUMMARY:
Patients with kidney failure on dialysis can be successfully transplanted. However, many of them do not attain a normal kidney function and/or present a slow deterioration of kidney function after transplantation. As a consequence, they can develop an endocrine disorder called hyperparathyroidism, which can cause bone disease and a high risk of bone fractures. In spite of the known bone disease and hyperparathyroidism, there is no well defined treatment for these patients.

Moreover, kidney transplant recipients present a higher mortality rate compared to the general population, and the principal cause of death is cardiovascular disease. Dialysis patients are known to have extensive cardiovascular calcifications and increased vascular stiffness, and these factors have been closely associated with cardiovascular mortality.

The effect of vitamin D on bone health is well known in the general population. Many studies showed a reduction in fracture rate in post-menopausal women and older men receiving vitamin D and calcium supplements. Vitamin D analogues are also commonly used to treat hyperparathyroidism in dialysis patients. Finally, vitamin D has been suggested to have beneficial effects on the cardiovascular system and to reduce mortality in dialysis patients.

Hectorol® is a vitamin D analog which has been demonstrated to effectively treat hyperparathyroidism in dialysis and pre-dialysis patients.

The effects of vitamin D supplementation on bone disease, hyperparathyroidism and cardiovascular function in kidney transplant recipients have not been properly studied.

Whether Hectorol® therapy helps reducing the severity of bone disease and improving vascular function in kidney transplant recipients is still unknown.

DETAILED DESCRIPTION:
The investigators plan to study the cardiovascular and bone effects of Hectorol® in 100 kidney transplant recipients. The kidney transplant patients will be screened for kidney transplant dysfunction and hyperparathyroidism. The study medication will be given to 50 patients. The other 50 patients will continue to be treated with the actual standard of care at the transplant clinic. Subjects will be followed for 18 months and their laboratory values, bone density, vascular calcification and stiffness will be collected to see if there is an effect of Hectorol® compared to the actual standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient > 18 year/old with reduced and stable kidney function (estimated GFR 25-60 ml/min/1.73m2)
* iPTH levels between 120 and 500 pg/ml
* Stable immunosuppressive therapy (5-10 mg Prednisone/day, stable dosage of calcineurin inhibitors, or other immunosuppressive agents for at least 6 months)

Exclusion Criteria:

* Recent rejection episode (< 3 months)
* One of the following: baseline estimated GFR>60 ml/min/1.73m2 or <25 ml/min/1.73m2, albumin-corrected Ca>9.5 mg/dl or serum phosphorus >4.6 mg/dl.
* Recipients of dual transplant organs with exception of kidney-pancreas
* Patients already receiving treatment with Vitamin D analogues
* Severe peripheral vascular disease or coronary artery disease
* History of previous parathyroidectomy
* Current alcohol or drug abuse
* Pregnant or nursing woman or female of child-bearing age not receiving contraception
* Other comorbidities that in the opinion of the investigators would reduce expected patient's survival and preclude study completion
* Medications that could interfere with Hectorol® metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Raggi and Antonio Guasch, MDs, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from July 2008 to February 2009
Pre-assignment Details: Four of the 12 subjects that were consented were withdrawn because they did not meet inclusion criteria or met exclusion criteria.
Groups:
- Doxercalciferol: Stable kidney transplant recipients will receive Doxercalciferol. The drug dosage will be initiated according to baseline iPTH levels. For patients with iPTH>300 pg/ml, oral Doxercalciferol will be given at 1 mcg/day; for patients with iPTH <300 pg/ml, oral Doxercalciferol will be initiated at 0.5 mcg/day.
- Control: Stable kidney transplant recipients do not receive any drug.
Period: Overall Study
Arm/Group | Doxercalciferol | Control
Started | 4 | 4
Completed | 0 | 0
Not Completed | 4 | 4
Not completed — Protocol terminated | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxercalciferol | Control | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With 50% Reduction of Intact Parathyroid Hormone (iPTH) Levels
Description: Number of participants that have 50% reduction in iPTH levels (but not lower than 65 pg/ml) at 18 months
Time Frame: 18 months
Population: Data not analyzed due to study termination
Arm/Group | Doxercalciferol | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Doxercalciferol | Control
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
Due to slow enrollment and primary investigator leaving institution, the study was terminated. Subjects were notified and those on active drug returned to their physicians to be treated according to standard of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes